CLINICAL TRIAL: NCT01648959
Title: Intra Cranial EEG Activity During Dexmedetomidine Sedation.Comparing the Effects of Dexmedetomidine on the Cortical and the Sub Cortical(Hippocampus) Structures.
Brief Title: Intra Cranial EEG Activity During Dexmedetomidine Sedation
Status: Terminated | Type: Observational
Why Stopped: Lack of funding
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Lashmi Venkatraghavan, Dr., University Health Network, Toronto
Other Study IDs: 12-0268
Record Dates: First submitted 2012-07-13; First posted 2012-07-25 (Estimated); Results first posted 2020-12-02 (Actual); Last update posted 2022-12-22 (Actual); Status verified 2022-12

CONDITIONS: Complex Partial Seizures
MeSH Terms: conditions — Seizures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: EEG Recording

SUMMARY:
Various parts of the brain are sensitive to various anesthetics.We like to study the effect of dexmedetomidine on the different parts of the brain in patients who are coming for DBS electrode removal under sedation.

DETAILED DESCRIPTION:
Cortical and sub cortical structures will have different sensitivities to various anesthetics.The objective of this study is to look at the changes in the intracranial electroencephalographic (EEG) characteristics during dexmedetomidine sedation and to determine the differences in the EEG characteristics between cortical and subcortical structures.

ELIGIBILITY:
Inclusion Criteria:

* Adults between 18 to 80 years of age, who are scheduled for elective removal of intracranial (surface and depth) electrodes under conscious sedation

Exclusion Criteria:

* Lack of informed consent
* Hypersensitivity to dexmedetomidine
* Language barrier
* Emergency surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults between 18 to 80 years of age, who are scheduled for elective removal of intracranial (surface and depth) electrodes under conscious sedation
Sampling Method: Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2012-07; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: lashmikumar venkatraghavan, MD, Principal Investigator — Assistant professor,Toronto western hospital,university health network (UHN)
Locations (1):
- Toronto Western Hospital,UHN., Toronto, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- iEEG Activity: iEEG data acquires every minute from the start of dexmedetomidine infusion to 5 minutes after the bolus dose.
Period: Overall Study
Arm/Group | iEEG Activity
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 5 patients who underwent elective removal of intracranial (neocortical and depth) electrodes under dexmedetomidine sedation were recruited for this prospective, non-randomized, observational study
Groups:
- Dexmedetomidine Infusion and iEEG Activity: 5 patients included in this study underwent bi-temporal implantation, and were shown to have unilateral hippocampal seizure onsets.
  iEEG data acquires every minute from the start of dexmedetomidine infusion to 5 minutes after the bolus dose.
Arm/Group | Dexmedetomidine Infusion and iEEG Activity
Number analyzed (Participants) | 5
Age, Customized [Mean (Standard Deviation); unit: years]
  Age | 37.3 (7.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 3
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: iEEG Recording
Description: iEEG data from each patient was analyzed using MATLAB (Natick, MA, USA). Data were presented as power spectral density, also referred to as the power spectrum or spectrum which quantifies the frequency distribution of energy or power within a signal. The spectrogram is a time-varying version of the spectrum. In these spectrograms, frequencies are arranged along the y-axis, and time along the x-axis, and power is indicated by color on a decibel (dB) scale. The power spectrum was computed for each channel using The Fast Fourier Transform (FFT). A window length of 20,000 data points was chosen in order to incorporate 4 cycles of a 1 Hz signal. The length of each window was therefore 4 seconds. A Hanning window was used to avoid edge effects of the windowing procedure. The length of the FFT was chosen to be 32768, which is the next power of 2 of the window length. The window overlap was set to zero.
Time Frame: 1 day
Measure: Mean (Full Range); unit: (Hz)
Groups:
- iEEG Activity: Data are presented as power spectral density, also referred to as the power spectrum or spectrum which quantifies the frequency distribution of energy or power within a signal.
Arm/Group | iEEG Activity
Number analyzed (Participants) | 5
(Hz) | 8 [0 to 10]

ADVERSE EVENTS:
Time Frame: From the time of induction to the end of surgical procedure
Description: No adverse events reported
Arm/Group | iEEG Activity
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes